CLINICAL TRIAL: NCT03026829
Title: "Cochlear Active Relief From Tinnitus (CART) Sound Therapy" for Tinnitus Relief in Nucleus® Cochlear Implant Users With Tinnitus
Brief Title: Sound Therapy for Tinnitus Relief in Cochlear Implant Users
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of subjects could not be achieved due to slow recruitment
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL5684
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Tinnitus, Hearing Loss, Cochlear Implant Users
Keywords: Sound therapy; Tinnitus relief
MeSH Terms: conditions — Tinnitus; Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART sound therapy (Experimental)
  Interventions: Device: CART sound therapy

INTERVENTIONS:
Device: CART sound therapy — The study consists of two parts:
  Phase 1: laboratory evaluation of CART sound acceptability
  Phase 2: take home evaluation of CART sound therapy including baseline without CART

SUMMARY:
The aim of this exploratory study is to evaluate the use and effectiveness of sound therapy for tinnitus relief in cochlear implant users with tinnitus. The sound therapy is a combination of tinnitus counselling and sound enrichment with the Cochlear Active Relief from Tinnitus (CART) firmware.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-reported tinnitus during standard Cochlear Implant (CI) activation for at least one month
* At least three months use of unilateral or bilateral Nucleus CI(s) driven by a CP900 Sound Processor. For bilateral use the most recently activated CI is used for at least three months
* Native speaker and fluency in the language used in the assessments (i.e. Dutch)

Exclusion Criteria:

* Additional handicaps that would prevent participation in evaluations
* History of psychiatric disorders or depression (on investigator's opinion)
* Unrealistic expectations as identified by the clinician on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the study
* Pulsatile or diagnosed objective / middle ear tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Quantification of Cochlear Implant (CI) patient's tinnitus via Visual Analogue Scale (VAS) | week 0
  Visual Analogue Scale (VAS) score on tinnitus
Quantification of Cochlear Implant (CI) patient's tinnitus via Visual Analogue Scale (VAS) | week 2
  Visual Analogue Scale (VAS) score on tinnitus
Quantification of Cochlear Implant (CI) patient's tinnitus via Visual Analogue Scale (VAS) | week 7
  Visual Analogue Scale (VAS) score on tinnitus
Quantification of Cochlear Implant (CI) patient's tinnitus via Tinnitus Functional Index (TFI) | week 0
Quantification of Cochlear Implant (CI) patient's tinnitus via Tinnitus Functional Index (TFI) | week 2
Quantification of Cochlear Implant (CI) patient's tinnitus via Tinnitus Functional Index (TFI) | week 7

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, PhD, Study Chair — Cochlear
Locations (2):
- Netherlands (2):
  - Department of Otorhinolaryngology, Maastricht University Medical Centre, Maastricht, Limburg
  - Department of Otorhinolaryngology, Head and Neck Surgery, Utrecht

REFERENCES:
- [Background] Tyler RS, Keiner AJ, Walker K, Deshpande AK, Witt S, Killian M, Ji H, Patrick J, Dillier N, van Dijk P, Lai WK, Hansen MR, Gantz B. A Series of Case Studies of Tinnitus Suppression With Mixed Background Stimuli in a Cochlear Implant. Am J Audiol. 2015 Sep;24(3):398-410. doi: 10.1044/2015_AJA-15-0005. PMID 26001407